CLINICAL TRIAL: NCT02207699
Title: Evaluation of the Effect of Benzonatate on QT Intervals Following Single Dose Administration of Benzonatate to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B3551003; BT-10-02
Record Dates: First submitted 2014-06-16; First posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — benzonatate; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Benzonatate 200 mg (Experimental)
  Interventions: Drug: Benzonatate 200 mg
- Benzonatate 800 mg (Experimental)
  Interventions: Drug: Benzonatate 800 mg
- Moxifloxacin 400 mg (Active Comparator)
  Interventions: Drug: Moxifloxacin 400 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benzonatate 200 mg — 2 benzonatate 100 mg perles and 6 placebo perles give by mouth once
  Arms: Benzonatate 200 mg
Drug: Benzonatate 800 mg — 8 benzonatate 100 mg perles given by mouth once
  Arms: Benzonatate 800 mg
Drug: Moxifloxacin 400 mg — 1 moxifloxacin 400 mg tablet given by mouth once
  Arms: Moxifloxacin 400 mg
Drug: Placebo — 8 placebo perles given by mouth once
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the effects of benzonatate (200 mg and 800 mg) on the QT interval following single dose oral administration at each time point post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12- lead ECG and clinical laboratory tests.
* Female subjects of non-childbearing potential must meet at least one of the following criteria:

  1. Achieved postmenopausal status, defined as: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum FSH level within the laboratory's reference range for postmenopausal females;
  2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
  3. Have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations and females that do NOT have a documented hysterectomy, bilateral oophorectomy and/or ovarian failure) will be considered to be of childbearing potential.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2, inclusive, and a total body weight >50 kg (110 lb).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all aspects of the study.
* Subjects willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Significant ECG abnormality at screening as determined by the investigator.
* History or risk factors of QT prolongation or torsades de pointes, congenital deafness and family history of sudden death.
* 12-lead ECG demonstrating QTcF >450 msec or a QRS interval >110 msec at Screening.
* Use of medications or dietary supplements capable of inducing or inhibiting hepatic enzyme metabolism or transport (e.g., barbiturates, rifampin, carbamazepine, phenytoin, primidone, or St. John's Wort) within 28 days of the first dose of study medication.
* Consumption of grapefruit or grapefruit containing products within 7 days prior to the first dose of study medication.
* Known history of hypersensitivity, allergy, severe adverse drug reaction or intolerance to quinolone antibiotics.
* Known hypersensitivity to benzonatate or other ester-type local anesthetics (ie, tetracaine, procaine).
* Subjects with a presence or history of dysphagia or difficulty swallowing pills.
* Subjects taking any concomitant anticonvulsant medications or with a history of seizure disorder.
* Subjects with a positive response to the question of actual attempt in the suicidal behavior section of the C-SSRS (Columbia-Suicide Severity Rating Scale). Subjects with active suicidal ideation with intent to act within 6 months of screening as determined by a positive response to questions 4 or 5 in the suicidal ideation section of the C-SSRS.
* Screening laboratory values considered clinically significant by the investigator.
* Screening supine blood pressure ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of rest.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Fridericia-corrected QTc change from the pre-dose time point to the post-dose time points following administration of study drug in therapeutic (200 mg) and supratherapeutic doses (800 mg). | -1, -0.75, -0.5, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 12, and 24 hours

SECONDARY OUTCOMES:
QT interval for Benzonatate, 4-(butylamino)benzoic acid (BBA-major metabolite of benzonatate), and moxifloxacin. | -1, -0.75, -0.5, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 12, and 24 hours
PR interval, QRS complex from single 12-lead electrocardiogram (ECG) | Screening, Day 0, and Day 1 at 4, 8, and 24 hours after dosing
Cmax (maximum plasma concentration) for BT and BBA measured in mcg/mL | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, and 12 hours
Tmax (time of maximum plasma concentration) for BT and BBA measured in minutes | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, and 12 hours
t½ (terminal half-life) for BT and BBA measured in minutes | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, and 12 hours
AUClast for BT and BBA measured in mcg•hr/mL | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, and 12 hours
AUCinf for BT and BBA measured in mcg•hr/mL | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, and 12 hours
Cmax(dn) for BT and BBA measured in mcg/mL | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, and 12 hours
AUClast(dn) for BT and BBA measured in mcg•hr/mL | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, and 12 hours
AUCinf(dn) for BT and BBA measured in mcg•hr/mL | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, and 12 hours
CL/F for BT measured in L/hr | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, and 12 hours
Vz/F for BT measured in L | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, and 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3551003&StudyName=Benzonatate%20QTc